CLINICAL TRIAL: NCT07393893
Title: The Effects of Parent-based IMPACT Intervention for Autism Sprectrum Disorder and Its Related Neural Mechanism
Brief Title: The Effects and Mechanism of Parent Intervention for Autism Sprectrum Disorder
Acronym: ImPACT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Weihua Zhao, Associate researcher, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UESTC-neuSCAN-101
Record Dates: First submitted 2025-12-10; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
Keywords: AUTISM; PARENT INTERVENTION; MECHANISM
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ImPACT-based Interventions (Experimental): Parent-based behavioral interventions for children.
  Interventions: Behavioral: Parents conducted interventions based on project ImPACT.
- General interventions (Active Comparator): Current routine interventions provided by behavioral trainers.
  Interventions: Behavioral: General behavioral interventions

INTERVENTIONS:
Behavioral: Parents conducted interventions based on project ImPACT. — Parents conduct behavioral interventions under the supervision of professional trainers who have obtained the certificate of Project IMPACT training. They are encouraged to conduct the interventions at least 10 hours per week without receiving other interventions from institutions or hospitals. Parents are asked to record the activities and duration of intervention they conducted daily in a logbook, which is reviewed weekly by certified trainers to ensure fidelity and provide feedback. Adherence is monitored through every other week one-one session to review progress, address challenges, and refine strategies. Trainers emphasize consistent implementation of evidence-based techniques, ensuring parents maintain high fidelity to the ImPACT model.
  Other Names: ImPACT
  Arms: ImPACT-based Interventions
Behavioral: General behavioral interventions — Children were subjected to interventions administered by behavioral trainers from hospitals or institutions. We advocated for them to persist with the existing interventions of any type (such as Applied Behavior Analysis, Discrete Trial Training, sensory integration, and language therapy) and augment the sessions to achieve a total of 10 hours per week, either in group or individual settings. Parents are asked to document the duration and type of sessions their children participated in each week in a notebook.
  Arms: General interventions

SUMMARY:
Purpose of the Research:

The goal of this clinical study is to investigate if a parent training program called "Project IMPACT" (Improving Parents as Communication Teachers) can help improve the core challenges in social interaction and communication for children with Autism Spectrum Disorder (ASD). And to explore whether and how this intervention affects children's brain activity.

Key Questions This Study Aims to Answer:

Does participation in the IMPACT parent training program significantly improve ASD symptoms, social communication abilities, and adaptive functioning in daily life for children with ASD compared to general intervention?

Study Design:

This is a assessor blinding randomized controlled trial. Participating children will be randomly assigned to one of two groups: IMPACT Intervention Group with primary caregiver conducting intervention and Control Group with current routine interventions provided by behavioral trainers.

The research team will evaluate all children at three time points: before the intervention starts, immediately after the 10 - week intervention period, and 6 months after the intervention ends. The measurements include social - related questionnaires, ADOS - 2, Griffiths Scales, eye - tracking, task - based fNIRS, and fMRI without sedation.

DETAILED DESCRIPTION:
Purpose of the Research:

The goal of this clinical study is to investigate if a parent training program called "Project IMPACT" (Improving Parents as Communication Teachers) can help improve the core challenges in social interaction and communication for children with Autism Spectrum Disorder (ASD). And to explore whether and how this intervention affects children's brain activity. We will use safe brain imaging techniques (such as MRI and functional Near-Infrared Spectroscopy, fNIRS) to compare changes in the brain before and after the intervention, aiming to understand the potential brain mechanisms behind behavioral progress. Ultimately, we hope to identify which types of children might benefit most from this intervention, providing insights for more personalized treatment recommendations in the future.

Key Questions This Study Aims to Answer:

Does participation in the IMPACT parent training program significantly improve ASD symptoms, social communication abilities, and adaptive functioning in daily life for children with ASD compared to general intervention?

Study Design:

This is a assessor blinding randomized controlled trial. Participating children will be randomly assigned to one of two groups:

IMPACT Intervention Group (approximately 40 children): The primary caregivers of these children will receive a systematic IMPACT training course over about 10 weeks (including group sessions and individual coaching), learning how to apply these techniques during interactions at home. All caregiver will be encouraged to conduct intervention at least 10 hours per week.

Control Group (approximately 40 children): The caregivers of these children will not receive IMPACT training during the initial 10-week period. They are encouraged to continue any current routine interventions their child is receiving. After 10 weeks, they will be offered the opportunity to receive the IMPACT training online for free as compensation.

Intervention Component (Exclusively for families randomly assigned to the ImPACT group):

Primary caregivers of participants will partake in the approximately 10 - week IMPACT parent training program. In weeks with odd numbers, caregivers will attend a group theory session lasting 3 - 4 hours. In weeks with even numbers, caregivers will receive a one - on - one coaching session (1 - 1.5 hours) with a trainer to enhance their intervention skills based on ImPACT. Caregivers are obligated to implement the learned strategies during daily home interactions with participants for a minimum of 10 hours per week and maintain a simple record of these activities. Trainers will monitor adherence via weekly reviews of activity logs and coaching sessions. Adherence will be further bolstered by real - time feedback during coaching sessions, where trainers prompt caregivers to engage their child in task - oriented activities while demonstrating and suggesting effective strategies, ensuring skill generalization in naturalistic settings.

The research team will evaluate all children at three time points: before the intervention starts, immediately after the 10-week intervention period, and 6 months after the intervention ends. The assessors will not know which group each child belongs to (they will be "blinded") to ensure objective results.

What the Involvement of Participation Entails:

If your child (aged 1.5 to 6.5 years) has a diagnosis of ASD and you agree to participate, the following may be involved:

Assessment Sessions (Three times: Pre-intervention, Post-intervention at 10 weeks, only SRS-2 measured after 6 months):

Questionnaires: You will be asked to fill out questionnaires about your child's behavior, social skills, and your own experiences and stress levels.

Child Assessments: A trained clinician, independent of the research team, will conduct standardized assessments of your child's development and social communication skills (e.g., ADOS-2, Griffiths Scales).

Eye-Tracking Test: Your child will watch short videos while a specialized, non-invasive device records where and for how long your child looks. This helps us understand their visual attention preferences towards social information.

Functional Near-Infrared Spectroscopy (fNIRS): During a play session, your child will wear a soft cap with sensors. It uses harmless near-infrared light to measure changes in brain activity in the outer layer of the brain. This procedure is safe, non-invasive, and radiation-free.

Magnetic Resonance Imaging (MRI) Scan (voluntary): We plan to conduct one brain MRI scan before and after the intervention for all willing participants to study brain structure and function. To ensure the child remains still during the scan, we plan to perform it during natural, deep sleep.

Voluntary Participation:

Participation in this study is completely voluntary. You may decide to withdraw yourself and your child from the study at any time, for any reason, without any penalty or effect on the future medical care you receive at this hospital or elsewhere.This study will be submitted for ethical review to ensure it meets scientific and ethical standards, protecting the rights, safety, and well-being of every participant.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 18 months and 78 months (6.5 years) at the time of enrollment.
* Participants must have received a formal diagnosis of autism spectrum disorder (or meet criteria for conditions within the autism spectrum) from qualified clinicians, such as psychiatrists or pediatricians, in accordance with the diagnostic criteria specified in either the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) or the International Classification of Diseases, 11th Revision (ICD-11).
* Participants must have a score meeting the autism spectrum cutoff on the Autism Diagnostic Observation Schedule, Second Edition (ADOS-2).
* At least one parent is able to participate in the entire assessment and intervention procedure.

Exclusion Criteria:

* Presence of a comorbid major neurological disorder (e.g., epilepsy, cerebral palsy) or a severe psychiatric condition.
* A history of significant brain injury or trauma.
* Current use of psychotropic medication or a within 3 months history of receiving transcranial electrical/magnetic stimulation therapy.
* Significant uncorrected impairment in visual or auditory acuity.
* Motor function disorders.

Ages: 18 Months to 78 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Autism Symptom Severity as measured by ADOS-2 Comparison Score and Subscales | From enrollment to the end of treatment at 10 weeks.
  The ADOS-2 (Autism Diagnostic Observation Schedule, Second Edition) is a semi-structured, standardized assessment of communication, social interaction, play, and restricted and repetitive behaviors. The Comparison Score is a standardized metric used to compare autism severity across different modules and ages. The Comparison Score ranges from 1 to 10, with higher scores indicating greater severity of autism spectrum-related symptoms (worse outcome).
Change in Social Impairment as measured by the Social Responsiveness Scale, Second Edition (SRS-2) Total Score | From enrollment to the end of treatment at 10 weeks, 3months after treatment.
  The SRS-2 is a 65-item caregiver-completed rating scale that measures the severity of autism spectrum symptoms as they occur in natural social settings. Each item is scored on a 4-point Likert scale ranging from 0 (Never True) to 3 (Almost Always True). The Total Raw Score is calculated by summing the scores of all 65 items. The total raw score ranges from 0 to 195, with higher scores indicating greater severity of social impairment (worse outcome).
Change in Child PFC Activation (Oxy-Hb) during Parent-Child Interaction | From enrollment to the end of treatment at 10 weeks.
  Mean Oxygenated Hemoglobin (Oxy-Hb) concentration in the Prefrontal Cortex (PFC) collected while the child engages in a standardized play task with their parent. Higher concentration indicates greater activation.
Change in Social Visual Preference Index (Percentage of Fixation Duration) | From enrollment to the end of treatment at 10 weeks.
  Participants view a battery of 3 paired paradigms presenting simultaneous social and non-social stimuli. The index is calculated as the percentage of total fixation duration spent on Social Areas of Interest (AOIs) divided by the total fixation duration on both Social and Non-social AOIs. Formula: (Duration on Social / (Duration on Social + Duration on Non-social)) * 100. The score is averaged across the 3 paradigms. Values range from 0 to 100%. Higher scores indicate a stronger preference for social stimuli.

SECONDARY OUTCOMES:
Change in Adaptive Functioning as measured by the ABAS-II General Adaptive Composite (GAC) and Domain Scores | From enrollment to the end of treatment at 10 weeks.
  The ABAS-II (Adaptive Behavior Assessment System, Second Edition) measures adaptive skills across the lifespan. It provides a General Adaptive Composite (GAC) score and three composite domain scores: Conceptual, Social, and Practical. These are reported as age-adjusted Standard Scores. The standard score range is 40 to 160 (Mean = 100, SD = 15). Unlike symptom scales, higher scores indicate better adaptive functioning (better outcome).
Change in Structural Brain Volume (Gray Matter Volume) in Regions of Interest (e.g., Prefrontal Cortex, Amygdala | From enrollment to the end of treatment at 10 weeks.
  Structural MRI data (T1-weighted) is collected during natural sleep. The metric reported is the Gray Matter Volume in specific Regions of Interest (ROIs) related to social processing.
  Data is preprocessed using standard pipelines (e.g., FreeSurfer). Values are reported in cubic millimeters ($mm^3$).
Change in Caregiver Burden as measured by the Caregiver Strain Questionnaire (CSQ) Total Score | From enrollment to the end of treatment at 10 weeks.
  The CSQ is a 21-item self-report measure used to assess the impact of caring for a child with emotional or behavioral disorders. It evaluates three domains: Objective Strain, Subjective Internalized Strain, and Subjective Externalized Strain. Items are rated on a 5-point scale ranging from 1 (Not at all a problem) to 5 (Very much a problem). The Total Score is calculated by summing the scores of all 21 items. The total score ranges from 21 to 105, with higher scores indicating higher levels of caregiver strain (worse outcome).
Change in Parenting Sense of Competence (PSOC): Total Score and Subscales | From enrollment to the end of treatment at 10 weeks.
  he PSOC is a 17-item self-report scale assessed on a 6-point Likert scale. It comprises two subscales: Satisfaction (9 items, reflecting the parent's motivation and frustration) and Efficacy (8 items, reflecting the parent's perceived competence and problem-solving ability). Items in the Satisfaction dimension are reverse-coded so that higher scores reflect greater satisfaction. The Total Score is the sum of all 17 items, ranging from 17 to 102. Subscale scores range from 9-54 (Satisfaction) and 8-48 (Efficacy). Higher scores indicate higher parenting self-esteem and better coping capability (better outcome).
Change in Repetitive Behaviors as measured by the Repetitive Behavior Scale-Revised (RBS-R) Total Score | From enrollment to the end of treatment at 10 weeks
  The RBS-R is a caregiver-rated questionnaire designed to measure the breadth and severity of repetitive behaviors in individuals with autism. It typically consists of 43 items grouped into six subscales (Stereotyped, Self-injurious, Compulsive, Ritualistic, Sameness, and Restricted Behavior). Each item is rated on a 4-point Likert scale ranging from 0 (Behavior does not occur) to 3 (Behavior occurs and is a severe problem). The Total Raw Score is the sum of all 43 items, ranging from 0 to 129. Higher scores indicate greater severity of repetitive behaviors (worse outcome).
Change in Social Communication Skills as measured by the Project ImPACT Social Communication Checklist (Parent-Reported) | From enrollment to the end of treatment at 10 weeks.
  he Social Communication Checklist is a psychometrically validated measure designed for the Project ImPACT intervention (Wainer, Berger, & Ingersoll, 2017). It assesses child progress across four domains: Social Engagement, Expressive Communication, Receptive Communication, and Imitation/Play. Items are scored on a frequency scale: 1 (Rarely/Not yet), 2 (Sometimes), and 3 (Frequently). (Note: Specific items 32-36 have weighted scoring for verbal/non-verbal strategies). The Total Score is the sum of all item scores, ranging from 70 to 215. Higher scores indicate better social communication skills (better outcome).
ADOS-2 Raw Scores (Module 1 and Module 2) | Baseline and Week 10
  Raw scores for the Social Affect (SA) and Restricted and Repetitive Behavior (RRB) domains, as well as the Overall Total Score. The specific algorithm (Module 1 "Few to No Words", Module 1 "Some Words", Module 2 "Younger than 5", or Module 2 "Older than 5") is determined by the participant's age and language level. Scores are summed, with higher scores indicating greater severity of autism spectrum-related symptoms (worse outcome). Scale Ranges: Social Affect (SA): 0 to 21, Restricted and Repetitive Behavior (RRB): 0 to 8, Total Score: 0 to 29 (Note: Maximum possible scores vary slightly by the specific algorithm used, but fall within these ranges.)
Change in Child PFC Activation (Oxy-Hb) during Interaction with Therapist | Baseline and Week 10
  Mean Oxy-Hb concentration in the PFC collected while the child plays with a therapist (unfamiliar adult). Used to assess generalization of social brain response.
Change in Child PFC Activation (Oxy-Hb) during Solitary Play | Baseline and Week 10
  Mean Oxy-Hb concentration in the PFC collected while the child plays alone (non-social condition). Serves as a control condition for social tasks.
Change in Social Orienting Index (Percentage of Fixation Counts) | Baseline and Week 10.
  Calculated as the percentage of discrete fixation counts directed towards Social AOIs relative to the total number of fixations on both stimuli types. Formula: (Count on Social / Total Count) * 100. Averaged across the 3 paradigms. Values range from 0 to 100%.
Change in Intrinsic Functional Connectivity (Resting State fMRI) | Baseline and Week 10
  Resting-state functional MRI is collected during natural sleep to assess intrinsic brain organization. The metric is the Functional Connectivity strength (Fisher's z-transformed correlation coefficient) within the Default Mode Network (DMN) or between social brain regions. Values range from -1 to 1 (approximate, after transformation). Higher values indicate stronger functional synchronization between regions.
Change in Parent Intervention Fidelity as measured by the Project ImPACT Fidelity of Implementation Rating Scale | Baseline and Week 10
  Assessed in the intervention group only.Parent fidelity is assessed by trained independent observers using the Project ImPACT Fidelity Checklist. The scale evaluates the parent's competence in five intervention domains: 1) Focus on the Child, 2) Adjust Communication, 3) Create Opportunities, 4) Teach New Skills, and 5) Shape the Interaction. Each domain is rated on a 5-point Likert scale ranging from 1 (Low Fidelity/Ineffective) to 5 (High Fidelity/Effective). The Total Score is reported as the Mean Score across all applicable items/domains. The range is 1 to 5. Higher scores indicate higher fidelity and competence in delivering the intervention (better outcome).
Change in Social Communication Skills as measured by the Project ImPACT Social Communication Checklist (Teacher/Coach-Reported) | Baseline and Week 10
  Assessed for the intervention group only. Completed by the teacher/interventionist to validate skill acquisition for the Project ImPACT intervention.It assesses child progress across four domains: Social Engagement, Expressive Communication, Receptive Communication, and Imitation/Play. Items are scored on a frequency scale: 1 (Rarely/Not yet), 2 (Sometimes), and 3 (Frequently). (Note: Specific items 32-36 have weighted scoring for verbal/non-verbal strategies). The Total Score is the sum of all item scores, ranging from 70 to 215. Higher scores indicate better social communication skills (better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu women's and children's central hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No